CLINICAL TRIAL: NCT06237062
Title: Real-world Experience of Patients Newly Started on Erenumab in the Gulf Region: a Longitudinal Prospective Observational Study
Brief Title: Migraine Survey in Gulf Region
Status: Terminated | Type: Observational
Why Stopped: Company decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAMG334AAE02
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Migraine
Keywords: migraine; survey; Gulf
MeSH Terms: conditions — Migraine Disorders | interventions — erenumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- adult migraine patients: adult migraine patients across the 4 Gulf Countries (UAE, Qatar, Oman and Kuwait)
  Interventions: Other: erenumab

INTERVENTIONS:
Other: erenumab — This was an observational study, there was no treatment allocation. After fulfilling the inclusion criteria and signing the informed consent, patients were directed through a link to the full survey.

SUMMARY:
The objective of this study was to evaluate the effect of erenumab on medication-specific treatment satisfaction in patients who newly started on erenumab over 12 weeks

DETAILED DESCRIPTION:
This was a longitudinal prospective descriptive primary data collection using a 20 min online survey. Patients were selected by investigators (general neurologists, headache/migraine specialists) in primary care clinics and hospitals. After fulfilling the inclusion criteria, the patient were asked to sign an online informed consent. A 5 min screener followed after which the patient was directed through a link to the full survey. The duration of data collection was for 6 months since the start of survey rolling in each site across centers in the Gulf Region.

ELIGIBILITY:
Inclusion Criteria:

* EM& CM (with or without Medication Overuse Headache (MOH)) patients
* Newly Started on erenumab either 70 mg or 140 mg (first dose received within 1 month prior study enrollment and baseline endpoints collection)
* Ability to receive 3 monthly doses of erenumab.
* Age more than 18 years
* Males and Females
* Allowing the patients to be stable on 1 adjunctive migraine preventive medication (if present)
* Agreed to be included in the study and signed informed consent

Exclusion Criteria:

* Less than 18 years
* Age at onset of Migraine more than 50 years
* Any contraindications to the start of erenumab as per label
* Refusal to sign informed consent
* Inability to participate or restricted access to the online survey
* Enrolled in an interventional migraine-related study at the time of the study enrollement

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinics in centers and hospitals treating adult migraine patients across the 4 Gulf Countries
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2024-06-05 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2024-11-18 (Actual)

PRIMARY OUTCOMES:
Mean score in the Treatment Satisfaction Questionnaire for Erenumab (TSQM) overall satisfaction scale score version 1.4 | 12 weeks
  TSQM is used to measure the Patients' self-reported satisfaction or dissatisfaction with the study treatment. The TSQM version 1.4 domain scores range from 0 to 100 with higher scores representing a higher satisfaction on that domain.

SECONDARY OUTCOMES:
Mean score in TSQM version 1.4 effectiveness domain | Week 12
  TSQM is used to measure the Patients' self-reported satisfaction or dissatisfaction with the study treatment. The TSQM version 1.4 domain scores range from 0 to 100 with higher scores representing a higher satisfaction on that domain.
Mean score in TSQM version 1.4 convenience domain | Week 12
  TSQM is used to measure the Patients' self-reported satisfaction or dissatisfaction with the study treatment. The TSQM version 1.4 domain scores range from 0 to 100 with higher scores representing a higher satisfaction on that domain.
Mean score in TSQM version 1.4 side effects domain | Week 12
  TSQM is used to measure the Patients' self-reported satisfaction or dissatisfaction with the study treatment. The TSQM version 1.4 domain scores range from 0 to 100 with higher scores representing a higher satisfaction on that domain.
Mean change from baseline in the score of HIT-6 | Baseline, Week 12
  Headache Impact Test (HIT-6) is a short-form self-administered questionnaire based on the internet-HIT question pool. The HIT-6 was developed as a global measure of adverse headache impact to assess headache severity in the previous month and change in a patient's clinical status over a short period of time. Six items assess the frequency of pain severity, headaches limiting daily activity (household, work, school, and social). Each of the 6 questions is responded to using 1 of 5 response categories: "never," "rarely," "sometimes," "very often," or "always." The total HIT-6 score ranges from 36 to 78. Lower values represent better outcomes, therefore negative change denotes improvement.
Mean change from baseline in the score of MIDAS at week 12 | Baseline, Week 12
  Migraine Disability Assessment (MIDAS) Questionnaire was developed to assess headache-related disability with the aim of improving migraine care. Headache sufferers answer five questions, scoring the number of days, in the past 3 months of activity limitations due to migraine.
  The total MIDAS score is the sum of the days given as response to these five questions (MIDAS 1 to MIDAS 5). The total score ranges from 0 to 90 and is used to categorize patients in disability grades I to IV. A higher score means more severe disability, placing the patient in a higher disability grade.
Mean change from baseline in the score of WPAI | Baseline, Week 12
  The Work Productivity Activity Impairment (WPAI) questionnaire measures the amount of absence or presence for work attendance and daily work activity impairment. A higher score on the WPAI indicates greater impairment and loss of productivity.
Mean change from baseline in the Patients' Global Impression of Change (PGIC) scale | Baseline, Week 12
  The PGIC evaluates overall health status as perceived by the patient in a seven-point single-item scale ranging from 'very much worse' to 'very much improved'
Mean change from baseline in MMDs | Baseline, Week 12
  Monthly Migraine Days (MMD), describes the number of days in a month with migraine.
Mean change from baseline in MSMDs | Baseline, Week 12
  Migraine specific medication treatment days (MSMD), describes the number of days per month with the use of migraine specific treatment.
Mean change from baseline in MHDs | Baseline, Week 12
  monthly headache days (MHD), is the number of days per month with headache.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to study results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18380